CLINICAL TRIAL: NCT05422235
Title: Comparison of the Effects of Different Exercise Programs on Lower Extremity Distal Tissue Mechanics, Muscle Strength and Neuropathy Symptoms in Type 2 Diabetics with Peripheral Neuropathy
Brief Title: The Effects of Different Exercises on Tissue Mechanics, Strength and Neuropathy Symptoms in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Cansu Koltak, Principal Investigator, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETK00-2021-0195
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Foot; Peripheral Neuropathy with Type 2 Diabetes
Keywords: Diabetic foot; Peripheral Neuropathy with Type 2 Diabetes; Aerobic exercise; stiffness
MeSH Terms: conditions — Diabetic Foot | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: The physiotherapist who evaluated the individuals participating in the study and the physiotherapist who took the treatment will not be the same. in addition, an independent statistician will do the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Other): Subjects in this group will be asked to continue their routine medical treatment for 24 weeks.
  Interventions: Other: Routine Medical Treatment
- Aerobic Exercise (Experimental): In order to determine the exercise capacity of subjects, submaximal exercise test will be performed.Aerobic training will be done 3 days a week for 12 weeks. Subjects will be followed for 24 weeks.
  Interventions: Other: Routine Medical Treatment; Other: Aerobic Exercise
- Aerobic Exercise+ Foot-Related Exercises (Experimental): In addition to walking training specific to the subject in the 2nd group, special exercises will be given to the feet and ankles. These exercises will be aimed at stretching, strengthening, increasing sensory input. Treatment program will be done 3 days a week for 12 weeks. Participants will be followed for 24 weeks.
  Interventions: Other: Routine Medical Treatment; Other: Aerobic Exercise+ Foot-Related Exercise

INTERVENTIONS:
Other: Routine Medical Treatment — Subjects will continue their routine medical treatment.
Other: Aerobic Exercise — Symptom-limited peak heart rates of subjects will be determined using the modified Bruce Protocol. For aerobic training, subject will be carried out on the treadmill according to the results of exercise tests. Initially, 40-60% of the peak heart rate will be trained and progression will be made in subject training programs every 2 weeks. Training will consist of warm-up, main exercise and cool-down periods. Aerobic training will be done 3 days a week for 12 weeks. Subjects will be followed for 24 weeks. The room temperature will be fixed at 25°C in order to keep the impact of environmental factors at a minimum. In addition, individuals will be asked to come with appropriate shoes and clothes for the training.
  Arms: Aerobic Exercise
Other: Aerobic Exercise+ Foot-Related Exercise — In addition to walking training specific to the subject in the aerobic exercise group, special exercises will be given to the feet and ankles. These exercises will be aimed at stretching, strengthening, increasing sensory input. Treatment program will be done 3 days a week for 12 weeks. Subjects will be followed for 24 weeks.
  Arms: Aerobic Exercise+ Foot-Related Exercises

SUMMARY:
To examine the effects of aerobic exercise and foot exercises in addition to aerobic exercise on lower extremity distal tissue mechanics, muscle strength and neuropathy symptoms in type 2 diabetics with peripheral neuropathy. Subjects will be divided into three groups through randomization.Subjects in the 1st group will be included in the control group and will continue their routine medical treatment for 12 weeks. Subjects in the 2nd group, in addition to their medical treatment, only aerobic exercise training,subjects in the 3rd group will be given aerobic exercise training and exercises for the foot and ankle in addition to their medical treatment. After 12 weeks of training, subjects will be followed for another 12 weeks. subjects will be evaluated before treatment, at 12 and 24 weeks.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is a chronic metabolic disease that causes fat, protein and carbohydrate metabolism disorders, characterized by hyperglycemia resulting from impaired insulin secretion and insulin activity or both of these factors. The "Sixth Diabetes Atlas" published by IDF (International Diabetes Federation) in 2013 contains important data about the current situation and future of diabetes in the world.Diabetic foot ulcer is shown as the reason for 15-20% of all diabetic individuals to apply to the hospital at least once. Diabetic foot is seen as a public health factor that increases the cost, as it increases the length of stay in the hospital, long-term antibiotic therapy, and overtime of many clinics such as surgery and orthopedics.

Musculoskeletal complications of diabetes are quite common. The severity of macrovascular and microvascular complications increases over time. It poses a risk for the formation of diabetic foot ulcers in diabetic individuals. It has been reported that joint mobility decreases in individuals, especially when the first metatarsophalangeal joint extension falls below 45 degrees, the risk increases. Decrease in distal muscle strength and atrophy occur due to peripheral neuropathy and axonal loss. Loss of strength causes various deformities in the foot. In addition, it has been stated that the plantar flexors are shortened and shortening increases the forefoot pressure in individuals with diabetes. A plantar pressure of more than 70 N/cm2 in the forefoot has also been reported as a risk factor for diabetic foot ulcer.

Physiotherapy approaches for symptoms should be applied in order to eliminate the risks of the disease and increase the quality of life after complications develop and their symptoms appear. Physiotherapy approaches are applied in primary, secondary and tertiary prevention. It is the duty of physiotherapists to educate the patient in primary prevention, to apply the most appropriate exercise training to prevent the development of diabetes-related complications in secondary prevention, and to apply the most appropriate physiotherapy approaches for diabetic foot and its treatment in tertiary prevention.

An important part of diabetic foot preventive methods is preventive exercise training.

Diabetic foot protective exercise aims to minimize the risks that occur or may occur.

Studies have reported that increased forefoot pressure is associated with decreased plantar fascia and Achilles flexibility. It has been stated that aerobic and resistance exercises are effective in glycemic control and HbA1c control, and the risk and symptoms of neuropathy are reduced. Contrary to popular belief, activities that involve standing do not increase the risk of ulceration. When the studies were examined, many studies were found that investigated the effects of aerobic exercise training and exercise training for the foot-ankle on normal joint range of motion, flexibility, muscle strength, walking speed and plantar pressure. However, no study has been found examining the effect of aerobic exercise training and exercise training for the foot and ankle on tissue stiffness.

Hypotheses:

H1: The effects of different exercise programs on lower extremity distal tissue mechanics are different in type 2 diabetics with peripheral neuropathy.

H2: The effects of different exercise programs on lower extremity distal muscle strength are different in type 2 diabetics with peripheral neuropathy.

H3: The effects of different exercise programs on neuropathy symptoms are different in type 2 diabetics with peripheral neuropathy.

H4: The effects of different exercise programs on plantar pressure are different in type 2 diabetics with peripheral neuropathy.

Material and Method:

The study will be conducted on subjects diagnosed with chronic mechanical type 2 diabetes due to distal peripheral neuropathy by specialist physician.Subjects who meet the inclusion and exclusion criteria and sign the informed consent form will be randomly divided into three different groups by random allocation program.

According to the power analysis made using the G-Power program; Assuming that the nonparametric ANOVA test will be used for the comparison between the 3 groups, a two-legged hypothesis will be established and a total of 93 people will be included in the calculation made by taking Cohen d=0.40, α=0.05, β=0.20, 31 in each group. It was decided to take 111 people from the research by predicting a 20% loss.

Subjects will be divided into three groups through randomization. Randomization will be done with random allocation software program. All groups will continue their routine medical treatments. All participants will be given subjects insoles and will be asked to use them for 24 weeks. Subjects in group 1 will continue their routine medical treatment for 12 weeks and will use insoles. Subjects in the 2nd group will be given only aerobic exercise training in addition to medical treatment and insoles, and the Subjects in the 3rd group will be given additional foot-ankle exercises for the 2nd group. Exercise training will continue for 12 weeks. For aerobic exercise training, Subjects will be walked on the treadmill three times a week. After the walking training, the Participants in the 3rd group will be given foot-ankle exercises. After 12 weeks of training, subjects will be followed for another 12 weeks. Participants will be evaluated before treatment, at 12 and 24 weeks. Evaluations and treatment will be done by different physical therapists. Physiotherapists making the assessment will not know which group the subjects are in.

Evaluations to be applied to the Subject:

Socio-demographic Form: In the first evaluation, socio-demographic information of subjects such as age, height, body weight will be obtained through a form. In addition to this information, the diabetes age of the subjects, the type of shoes used, the history of ulceration, the presence of other accompanying chronic diseases and their medications will be questioned.

Physical activity levels: It will be evaluated with the SenseWear Armband (SWA). Individuals will be asked to use two days a week and one day on the weekend. They will be asked to remove the device only while bathing. It is a small and lightweight device to be placed at the midpoint of the triceps muscle on the right arm. It has been developed to measure energy consumption more accurately by combining biaxial accelerometer and physical parameters. It includes motion and temperature sensors. It consists of biaxial accelerometer, skin temperature sensor, galvanic skin response and heat flux sensor. Body surface temperature will be evaluated with the skin temperature sensor, and skin impedance, which reflects the water content of the skin and the construction and dilatation of the vascular periphery, will be evaluated with the Galvanic Skin Response sensor. In addition, the rate of heat dissipation from the body will be evaluated with the Heat Flux Sensor, and the motion will be evaluated with the biaxial accelerometer. With the help of the program, personal information is entered on the screen, the calories consumed, the value in MET, the number of steps, rest, supine position and physical activity.

Evaluation of Foot Postures: Foot posture will be assessed by the Foot Posture Index (FPI).

Light Touch Pressure Sense Assessment: Plantar light touch-pressure sense is derived from 9 regions of Semmes-Weinstein® type (Baseline® Tactile), including heel, medial midfoot, lateral midfoot, 1st, 3rd and 5th metatarsal head and 1st, 3rd and 5th fingers. The Sensory Evaluator will be evaluated using 6 different monofilaments (levels: 2.83; 3.61; 4.31; 4.56; 5.07; 6.65), each of equal length (38 mm) and different diameters, applying standard pressure to the skin.

Blood values: Plasma glucose level, HbA1c, B 12, Urinary Albumin, CRP values will be taken in the medical analysis laboratory.

Neuropathy symptoms will be evaluated with the Douleur Neuropathique 4, Lanss Pain questionnaire.

Vibration test: Vibration sense will be evaluated quantitatively with a biotesiometer.

Stiffness assessment: It will be evaluated in continuous passive motion mode using an isokinetic dynamometer device (Humac Norm Isocynetic Dynanometer).

Plantar-Dorsiflexion Muscle Strength: Strength values of isokinetic ankle plantar flexor and dorsiflexor muscles will be measured by using an isokinetic dynamometer device (Humac Norm Isocynetic Dynanometer).

Plantar Pressure: Plantar pressures will be evaluated with a fixed pedobarograph (Medilogic, platform basic; Germany) and a 2-step protocol. Measurements will be recorded barefoot and for both feet separately. The sole of the foot will be divided into 10 regions (thumb, other fingers, 1st metatarsal head, 2nd metatarsal head, 3rd metatarsal head, 4th metatarsal head, 5th metatarsal head, lateral foot, medial and lateral heel). The peak pressure (N/cm2) in each zone will be noted.

Evaluation of foot function: Foot function will be evaluated using the Turkish version of the Foot Function Index (FFI). This questionnaire, which is used in foot and ankle problems, consists of 3 sub-headings and 23 items: foot pain level, disability and activity limitation.

Quality of life assessment: Turkish version of Nottingham Health Profile will be used.

All assessments will be made before treatment, at week 12, and week 24.

Interventions:

1. Group: Subjects will continue their routine medical treatments and will use custom made insoles for 24 weeks.
2. Group (Aerobic Exercises): Subjects will continue their routine medical treatments and will use custom made insoles for 24 weeks. In order to determine the exercise capacity of individuals, submaximal exercise test will be performed. Symptom-limited peak heart rates of individuals will be determined using the modified Bruce Protocol. For aerobic training, individuals will be carried out on the treadmill according to the results of exercise tests. Initially, 40-60% of the peak heart rate will be trained and progression will be made in individual training programs every 2 weeks. Aerobic exercise will be done for 12 weeks, 3 days a week. Walking will be done for aerobic exercise. The room temperature will be fixed at 25°C in order to keep the impact of environmental factors at a minimum. In addition, individuals will be asked to come with appropriate shoes and clothes for the training.
3. Group (Aerobic exercises+ Foot-related exercises): In addition to group 2, exercises that will increase the stretching, strengthening and sensory input for the ankles of the subjects will be given. Exercises for the foot and ankle will be done after the aerobic exercise is over. Aerobic exercise and foot related exercises will be done for 12 weeks, 3 days a week. Walking will be done for aerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Type 2 DM
* Being able to walk independently
* Getting at least 23 points from the mini mental test
* Patients with peripheral neuropathy according to ADA criteria

Exclusion Criteria:

* Presence of active ulcer
* Amputation history
* History of lower extremity surgery
* Participating in a regular exercise program in the last three months
* Having a Charcot deformity
* Presence of major vascular complications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Changes passive ankle stiffness compared with baseline and last measurement and Follow-up | Subjects will be evaluated before treatment, at week 12, and week 24. The assessment takes approximately 20 minutes.
  Passive ankle stiffness will be measured before treatment, after treatment, and at follow-up.passive ankle stiffness will be evaluated with an isokinetic dynamometer.

SECONDARY OUTCOMES:
Changes Plantar Flexion and Dorsiflexion muscle strength compared with baseline and last measurement and Follow-up | Subjects will be evaluated before treatment, at week 12, and week 24. The assessment takes approximately 20 minutes.
  Plantar Flexion and Dorsiflexion strength will be evaluated concentrically with isokinetic dynamometer.
Changes Douleur Neuropathique 4 (DN4) compared with baseline and last measurement and Follow-up | Subjects will be evaluated before treatment, at week 12, and week 24. The assessment takes approximately 10 minutes.
  Neuropathy symptoms will be assessed using the Douleur Neuropathique.Neuropathic pain will be evaluated with the Douleur Neuropathique 4 (DN4) Pain diagnostic questionnaire. The questionnaire contains 10 items, 3 of which are related to the neurological examination. Questionnaire; He questions the symptoms of burning, painful cold sensation, electric shock sensation, tingling, prickling, numbness and itching. Neurological examination includes light touch hypoesthesia, needle prick hypoesthesia, and brushing allodynia. Each question with a yes answer is awarded 1 point. The maximum score to be obtained with the sum of the symptoms and clinical examination is 10. The Turkish validity and reliability was determined by Çevik et al., and it was defined as neuropathic pain with a sensitivity of 95% and a specificity of 96.6% with a score of 4 and above.
Changes plantar pressure compared with baseline and last measurement and Follow-up | Subjects will be evaluated before treatment, at week 12, and week 24. The assessment takes approximately 10 minutes.
  Plantar pressures will be evaluated with a fixed pedobarograph (Medilogic, platform basic; Germany) and a 2-step protocol.
Changes foot function compared with baseline and last measurement and Follow-up | Subjects will be evaluated before treatment, at week 12, and week 24. The assessment takes approximately 5 minutes.
  Foot function will be evaluted with Turkısh version Foot Function Index (FFI). This questionnaire, which is used in foot and ankle problems, consists of 3 sub-headings and 23 items: foot pain level, disability and activity limitation. 9 items question foot pain severity, 9 items insufficiency level, 5 items activity limitation.
  FFI is a valid and reliable scale, with each item scored between 0 and 10 according to the visual analog scale, by the individual himself. The higher the FFI score, the more pain, disability, and activity limitation are interpreted.
Changes quality of life compared with baseline and last measurement and Follow-up | Subjects will be evaluated before treatment, at week 12, and week 24. The assessment takes approximately 5 minutes.
  Quality of Life will be evulated with Turkish version Nottingham Health Profile (NHP). NHP is a general quality of life questionnaire that measures the perceived health problems of the individual and the extent to which these problems affect normal daily activities. The questionnaire consists of 38 items and evaluates six dimensions related to health status: Energy (3 items), pain (8 items), emotional reactions (9 items), sleep (5 items), social isolation (5 items), and physical activity (8 items). matter). Questions are answered with yes or no. Each section is scored between 0-100. 0 indicates best health, 100 indicates worst health.
Changes (Leeds Assesment of Neuropathic Symptoms and Signs (LANSS) compared with baseline and last measurement and Follow-up | Subjects will be evaluated before treatment, at week 12, and week 24. The assessment takes approximately 10 minutes.
  Neuropathy symptoms will be assessed using the LANSS. LANSS consists of two parts; The first part, filled in by the patient, and the second part, which includes a brief physical examination of the investigator. With five questions (max16 points) answered by the patient himself, his experiences related to neuropathic pain are described. In the physical examination part, the presence of allodynia is tested by touching the painful and painless area with cotton. In addition, the perception of pinprick is evaluated in the same areas by using a 23-gauge needle. With the verbal description of the person and the score obtained as a result of the neurological examination, it is decided that the patient's pain is neuropathic or nociceptive in character. A score of 12 and above is classified as neuropathic, and below 12 as nociceptive pain.
Changes Michigan Neuropathy Screening Instrument (MSNI) compared with baseline and last measurement and Follow-up | Subjects will be evaluated before treatment, at week 12, and week 24. The assessment takes approximately 10 minutes.
  Neuropathy symptoms will be assessed using the MSNI. MSNI consists of two parts. The first part, consisting of 15 questions, evaluates pain, numbness and temperature sensitivity. Questions are answered with yes or no. The maximum score is 13, indicating the presence of more neuropathic symptoms as the score increases. In the second part, those who score 2 or more out of 10 points are considered to have neuropathy.The second part of the MSNI includes a brief physical assessment by healthcare professionals. There are 5 titles in total to be evaluated separately for the right and left feet.
Changes vibration test compared with baseline and last measurement and Follow-up | Subjects will be evaluated before treatment, at week 12, and week 24. The assessment takes approximately 15 minutes.
  Vibration sense will be evaluated quantitatively with a biotesiometer. Vibration sense will be evaluated quantitatively with a biotesiometer. The measurement will be made by applying a probe to the thumb. The probe will vibrate to the region of increasing intensity and the point at which the patient feels the vibration will be accepted as the measurement threshold. The biotesiometer can show values between 0-50 volts. Individuals with a vibration detection threshold above 25 Volts will be considered to have neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Cansu KOLTAK, MSc, Principal Investigator — Eastern Mediterranean University; Yasin YURT, PhD, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Mersin, Famagusta, Turkey (Türkiye)

REFERENCES:
- [Background] Diabetes Canada Clinical Practice Guidelines Expert Committee; Punthakee Z, Goldenberg R, Katz P. Definition, Classification and Diagnosis of Diabetes, Prediabetes and Metabolic Syndrome. Can J Diabetes. 2018 Apr;42 Suppl 1:S10-S15. doi: 10.1016/j.jcjd.2017.10.003. No abstract available. PMID 29650080
- [Background] Spijkerman AM, Dekker JM, Nijpels G, Adriaanse MC, Kostense PJ, Ruwaard D, Stehouwer CD, Bouter LM, Heine RJ. Microvascular complications at time of diagnosis of type 2 diabetes are similar among diabetic patients detected by targeted screening and patients newly diagnosed in general practice: the hoorn screening study. Diabetes Care. 2003 Sep;26(9):2604-8. doi: 10.2337/diacare.26.9.2604. PMID 12941726
- [Background] Amos AF, McCarty DJ, Zimmet P. The rising global burden of diabetes and its complications: estimates and projections to the year 2010. Diabet Med. 1997;14 Suppl 5:S1-85. PMID 9450510
- [Background] Raghav A, Khan ZA, Labala RK, Ahmad J, Noor S, Mishra BK. Financial burden of diabetic foot ulcers to world: a progressive topic to discuss always. Ther Adv Endocrinol Metab. 2018 Jan;9(1):29-31. doi: 10.1177/2042018817744513. Epub 2017 Dec 12. PMID 29344337
- [Background] Brownrigg JR, Apelqvist J, Bakker K, Schaper NC, Hinchliffe RJ. Evidence-based management of PAD & the diabetic foot. Eur J Vasc Endovasc Surg. 2013 Jun;45(6):673-81. doi: 10.1016/j.ejvs.2013.02.014. Epub 2013 Mar 27. PMID 23540807
- [Background] Allet L, Armand S, de Bie RA, Golay A, Monnin D, Aminian K, Staal JB, de Bruin ED. The gait and balance of patients with diabetes can be improved: a randomised controlled trial. Diabetologia. 2010 Mar;53(3):458-66. doi: 10.1007/s00125-009-1592-4. Epub 2009 Nov 17. PMID 19921145
- [Background] Lavery LA, Armstrong DG, Boulton AJ; Diabetex Research Group. Ankle equinus deformity and its relationship to high plantar pressure in a large population with diabetes mellitus. J Am Podiatr Med Assoc. 2002 Oct;92(9):479-82. doi: 10.7547/87507315-92-9-479. PMID 12381796
- [Background] Mueller MJ. People with diabetes: a population desperate for movement. Phys Ther. 2008 Nov;88(11):1250-3. doi: 10.2522/ptj.2008.88.11.1250. Epub 2008 Sep 18. No abstract available. PMID 18801849
- [Background] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Background] Mueller MJ, Tuttle LJ, Lemaster JW, Strube MJ, McGill JB, Hastings MK, Sinacore DR. Weight-bearing versus nonweight-bearing exercise for persons with diabetes and peripheral neuropathy: a randomized controlled trial. Arch Phys Med Rehabil. 2013 May;94(5):829-38. doi: 10.1016/j.apmr.2012.12.015. Epub 2012 Dec 28. PMID 23276801
- [Background] Heiermann S, Khalaj Hedayati K, Muller MJ, Dittmar M. Accuracy of a portable multisensor body monitor for predicting resting energy expenditure in older people: a comparison with indirect calorimetry. Gerontology. 2011;57(5):473-9. doi: 10.1159/000322109. Epub 2010 Dec 22. PMID 21196692
- [Background] Papazoglou D, Augello G, Tagliaferri M, Savia G, Marzullo P, Maltezos E, Liuzzi A. Evaluation of a multisensor armband in estimating energy expenditure in obese individuals. Obesity (Silver Spring). 2006 Dec;14(12):2217-23. doi: 10.1038/oby.2006.260. PMID 17189549
- [Background] Troosters T, Sciurba F, Battaglia S, Langer D, Valluri SR, Martino L, Benzo R, Andre D, Weisman I, Decramer M. Physical inactivity in patients with COPD, a controlled multi-center pilot-study. Respir Med. 2010 Jul;104(7):1005-11. doi: 10.1016/j.rmed.2010.01.012. Epub 2010 Feb 18. PMID 20167463
- [Background] Redmond AC, Crosbie J, Ouvrier RA. Development and validation of a novel rating system for scoring standing foot posture: the Foot Posture Index. Clin Biomech (Bristol). 2006 Jan;21(1):89-98. doi: 10.1016/j.clinbiomech.2005.08.002. Epub 2005 Sep 21. PMID 16182419
- [Background] Dros J, Wewerinke A, Bindels PJ, van Weert HC. Accuracy of monofilament testing to diagnose peripheral neuropathy: a systematic review. Ann Fam Med. 2009 Nov-Dec;7(6):555-8. doi: 10.1370/afm.1016. PMID 19901316
- [Background] Bouhassira D, Attal N, Alchaar H, Boureau F, Brochet B, Bruxelle J, Cunin G, Fermanian J, Ginies P, Grun-Overdyking A, Jafari-Schluep H, Lanteri-Minet M, Laurent B, Mick G, Serrie A, Valade D, Vicaut E. Comparison of pain syndromes associated with nervous or somatic lesions and development of a new neuropathic pain diagnostic questionnaire (DN4). Pain. 2005 Mar;114(1-2):29-36. doi: 10.1016/j.pain.2004.12.010. Epub 2005 Jan 26. PMID 15733628
- [Background] Unal-Cevik I, Sarioglu-Ay S, Evcik D. A comparison of the DN4 and LANSS questionnaires in the assessment of neuropathic pain: validity and reliability of the Turkish version of DN4. J Pain. 2010 Nov;11(11):1129-35. doi: 10.1016/j.jpain.2010.02.003. Epub 2010 Apr 24. PMID 20418179
- [Background] Yucel A, Senocak M, Kocasoy Orhan E, Cimen A, Ertas M. Results of the Leeds assessment of neuropathic symptoms and signs pain scale in Turkey: a validation study. J Pain. 2004 Oct;5(8):427-32. doi: 10.1016/j.jpain.2004.07.001. PMID 15501424
- [Background] Karvestedt L, Martensson E, Grill V, Elofsson S, von Wendt G, Hamsten A, Brismar K. Peripheral sensory neuropathy associates with micro- or macroangiopathy: results from a population-based study of type 2 diabetic patients in Sweden. Diabetes Care. 2009 Feb;32(2):317-22. doi: 10.2337/dc08-1250. Epub 2008 Nov 25. PMID 19033412
- [Background] Woodson C, Bandy WD, Curis D, Baldwin D. Relationship of isokinetic peak torque with work and power for ankle plantar flexion and dorsiflexion. J Orthop Sports Phys Ther. 1995 Sep;22(3):113-5. doi: 10.2519/jospt.1995.22.3.113. PMID 8535468
- [Background] Bus SA, de Lange A. A comparison of the 1-step, 2-step, and 3-step protocols for obtaining barefoot plantar pressure data in the diabetic neuropathic foot. Clin Biomech (Bristol). 2005 Nov;20(9):892-9. doi: 10.1016/j.clinbiomech.2005.05.004. PMID 15996799
- [Background] Lobmann R, Kayser R, Kasten G, Kasten U, Kluge K, Neumann W, Lehnert H. Effects of preventative footwear on foot pressure as determined by pedobarography in diabetic patients: a prospective study. Diabet Med. 2001 Apr;18(4):314-9. doi: 10.1046/j.1464-5491.2001.00482.x. PMID 11437863
- [Background] Budiman-Mak E, Conrad KJ, Mazza J, Stuck RM. A review of the foot function index and the foot function index - revised. J Foot Ankle Res. 2013 Feb 1;6(1):5. doi: 10.1186/1757-1146-6-5. PMID 23369667
- [Background] Noonan V, Dean E. Submaximal exercise testing: clinical application and interpretation. Phys Ther. 2000 Aug;80(8):782-807. PMID 10911416